CLINICAL TRIAL: NCT00202384
Title: Gene Expression in MS Patients Before and During Treatment With High-dose Interferon Beta: Prospective Study for the Identification of Predicting Factors of Therapeutic Response.
Brief Title: Gene Expression in MS Patients Before and During Treatment With Interferon-beta
Status: Terminated | Type: Observational
Why Stopped: Few participants enrolled
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Ristori, MD, S. Andrea Hospital
Other Study IDs: NEU - FCG - 02
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; microarrays
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinical and experimental evidences suggest that there is a variability in therapeutic response to immunomodulating therapies in Multiple Sclerosis patients.

Microarrays is a technology that permits to monitor the expression levels of thousands of genes at a time.

The specific aim of this study is to identify predictive factors of therapeutic response in MS patients treated with high-dose Interferon-Beta.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsing-remitting MS (McDonald criteria)
* age between 18-55
* EDSS less or equal to 5.5

Exclusion Criteria:

* use of any other disease modifying drugs
* use of corticosteroids during 3 months before starting protocol
* clinical relapse during 1 month before starting protocol
* serious heart, renal, hepatic or haematological dysfunction defined by laboratory exams

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Outpatient MS centres
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2004-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Gene Expression in MS Patients | baseline and 12 months after IFN beta 1a treatment
  Change in Gene Expression profile in MS Patients at 12 months of IFN beta 1a treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marco Salvetti, MD, Study Director
Locations (1):
- Azienda Ospedaliera S. Andrea, II Facoltà di Medicina e Chirurgia, Università di Roma "La Sapienza", Rome, Italy

REFERENCES:
- [Background] Bomprezzi R, Ringner M, Kim S, Bittner ML, Khan J, Chen Y, Elkahloun A, Yu A, Bielekova B, Meltzer PS, Martin R, McFarland HF, Trent JM. Gene expression profile in multiple sclerosis patients and healthy controls: identifying pathways relevant to disease. Hum Mol Genet. 2003 Sep 1;12(17):2191-9. doi: 10.1093/hmg/ddg221. Epub 2003 Jul 8. PMID 12915464
- [Background] Sturzebecher S, Wandinger KP, Rosenwald A, Sathyamoorthy M, Tzou A, Mattar P, Frank JA, Staudt L, Martin R, McFarland HF. Expression profiling identifies responder and non-responder phenotypes to interferon-beta in multiple sclerosis. Brain. 2003 Jun;126(Pt 6):1419-29. doi: 10.1093/brain/awg147. PMID 12764062
- [Background] Weinstock-Guttman B, Badgett D, Patrick K, Hartrich L, Santos R, Hall D, Baier M, Feichter J, Ramanathan M. Genomic effects of IFN-beta in multiple sclerosis patients. J Immunol. 2003 Sep 1;171(5):2694-702. doi: 10.4049/jimmunol.171.5.2694. PMID 12928423
- [Background] Waubant E, Vukusic S, Gignoux L, Dubief FD, Achiti I, Blanc S, Renoux C, Confavreux C. Clinical characteristics of responders to interferon therapy for relapsing MS. Neurology. 2003 Jul 22;61(2):184-9. doi: 10.1212/01.wnl.0000078888.07196.0b. PMID 12874396